CLINICAL TRIAL: NCT02428660
Title: Medication Therapy Management Combined With Drug and Gene Interaction Software and Cytochrome DNA Testing Among a Population of Polypharmacy Medicare Patients
Brief Title: Drug & Gene Interaction Risk Analysis With & Without Genetic Testing Among Patients Undergoing MTM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Genelex Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: Genelex 2014-02
Record Dates: First submitted 2015-04-21; First posted 2015-04-29 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Cytochrome P450 CYP2D6 Enzyme Deficiency; Poor Metabolizer Due to Cytochrome P450 CYP2D6 Variant; Ultrarapid Metabolizer Due to Cytochrome P450 CYP2D6 Variant; Extensive Metabolizer Due to Cytochrome P450 CYP2D6 Variant; Cytochrome P450 CYP2C9 Enzyme Deficiency; Cytochrome P450 CYP2C19 Enzyme Deficiency; Drug Metabolism, Poor, CYP2D6-RELATED; Drug Metabolism, Poor, CYP2C19-RELATED; CYP2D6 Polymorphism
Keywords: Polypharmacy; Chronic conditions; Drug Therapy Problems; Medication Therapy Management; Medication-Related Problems; CYP3A4; CYP3A5; Drug-drug interactions; Drug-gene interactions; Drug-drug-gene interactions; Adverse Drug Reactions; Activities of Daily Living
MeSH Terms: conditions — Drug Metabolism, Poor, CYP2D6-Related; Drug Metabolism, Poor, CYP2C19-Related; Chronic Disease; Drug-Related Side Effects and Adverse Reactions | interventions — Pharmacogenomic Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Controls (no analysis or testing) (Other): MTM alone (i.e. Treatment As Usual)
  Interventions: Other: MTM
- Group 1 (Experimental): MTM + software-based drug & gene interaction risk analysis + pharmacogenetic testing
  Interventions: Genetic: Pharmacogenetic testing; Other: Software-based drug & gene interaction risk analysis; Other: MTM
- Group 2 (Active Comparator): MTM + software-based drug & gene interaction risk analysis only
  Interventions: Other: Software-based drug & gene interaction risk analysis; Other: MTM

INTERVENTIONS:
Genetic: Pharmacogenetic testing — Genetic testing for 2D6, 2C9, 2C19, 3A4, 3A5 polymorphisms
  Other Names: YouScript(R) Personalized Prescribing System
  Arms: Group 1
Other: Software-based drug & gene interaction risk analysis — By assessing a patient's medication list along with the frequencies of variant phenotypes in the population, YouScript is able to identify whether a patient might be at risk for an adverse drug event and suggest when testing might be appropriate.
  Arms: Group 1; Group 2
Other: MTM — Medication Therapy Management

SUMMARY:
This randomized controlled trial will evaluate whether the use of pharmacogenetic testing through a Medication Therapy Management (MTM) program has a beneficial impact on drug therapy problems. More specifically, cytochrome DNA testing, which provides information with regards to participant specific metabolism of medications, will be used in the evaluation of participant medication regimens. The overall aim of the project is to evaluate if the addition of genetic CYP testing to a standardized MTM Program provides increased clinical value. To answer this question, the investigators will look at the drug therapy problems (DTPs) identified by the genetic test compared to those DTPs discovered without the test.

DETAILED DESCRIPTION:
All study participants will receive a Comprehensive Medication Review (CMR). One third will have standard MTM conducted. Another third of the participants will be randomized to MTM plus drug interaction risk analysis via YouScript software. The remaining third will be randomized to MTM along with drug interaction risk analysis via YouScript software and genetic testing. The software will identify polypharmacy patients who may benefit from pharmacogenetic testing based on their current medication regimen. Results of the testing will be mailed to both the participant and their provider. Participants who undergo testing will also receive a follow-up phone call. All participants, including those who receive MTM alone, will receive a contact 3 months later to assess quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Aged 65 or over and enrolled in a Medicare Part-D Prescription Drug Plan.
* Currently prescribed ≥6 chronic medications.
* Have ≥3 chronic disease states including osteoarthritis, rheumatoid arthritis, heart failure, diabetes, dyslipidemia, hypertension, asthma, chronic obstructive pulmonary disease, atrial fibrillation, and coronary artery disease.
* Participant incurred the Medicare-mandated dollar amount in medication-related costs in the previous quarter.

Exclusion Criteria:

* Inability to perform MTM encounter due to living situation (e.g. patient is enrolled in hospice, or is in long term care facility).
* Patient is unable to perform MTM encounter due to metal health barriers as described by Brief Interview for Mental Status (BIMS) score of <13 points.
* Patient identifies themselves as being unable to perform the oral swab function of the genetic test.
* Patient had a known MTM session within the preceding 12 months.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 341 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Number of Drug Therapy Problems (DTPs) | Baseline
  Tabulation of the number of drug therapy problems identified by drug & gene interaction risk analysis, with and without genetic testing.

SECONDARY OUTCOMES:
Number of adverse drug reactions | 8 months
  Tabulation of adverse drug reactions.
Quality of Life | 3 months
  Assessment of quality of life score via SF-12.

OTHER OUTCOMES:
Acceptance of recommendations by pharmacists | Baseline
  Proportion of recommendations deemed clinically relevant by local pharmacists.
Major event risk reduction | 8 months
  Tabulation of major health events avoided (e.g. stroke, heart attack, and other events requiring hospitalization).
Acceptance of recommendations by clinician providers | 8 months
  Proportion of recommendations resulting in medication or dose changes.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan W Magness, PharmD, Principal Investigator — VRx Pharmacy Services
Locations (1):
- VRx Pharmacy Services, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kim K, Magness JW, Nelson R, Baron V, Brixner DI. Clinical Utility of Pharmacogenetic Testing and a Clinical Decision Support Tool to Enhance the Identification of Drug Therapy Problems Through Medication Therapy Management in Polypharmacy Patients. J Manag Care Spec Pharm. 2018 Dec;24(12):1250-1259. doi: 10.18553/jmcp.2018.24.12.1250. PMID 30479202
- See also: Demo of YouScript(R) Personalized Prescribing System — http://youscript.com/demo/